CLINICAL TRIAL: NCT05966376
Title: Efficacy and Safety of Hemostatic Methods in Distal Radial Artery Approach for Cardiac Catheterization
Acronym: HEMOSTAD-INC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Arnoldo Enmanuel Loáisiga Sáenz, Interventional Cardiology, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-1255
Record Dates: First submitted 2023-04-05; First posted 2023-07-28 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Coronary Intervention; Transradial Approach
Keywords: Distal Radial Artery Access; PreludeSYNC distal; Terumo Radial Band

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified Terumo Radial Band (Experimental): A standard hemostatic device used for proximal radial approach. The hard plastic component is removed to achieve better attachment in the distal radial approach.
  * Clean and dry the puncture site.
  * The introducer is withdrawn 2 cm.
  * Place the device on the patient's hand depending on the approach side.
  * Terumo logo is positioned toward the little finger side.
  * The green mark is positioned 1 cm proximal to the puncture site.
  * The bands are adjusted and fixed around the wrist.
  * The Terumo syringe is filled with 15 ml of air.
  * The balloon of the device is slowly inflated through the valve while the introducer is slowly withdrawn simultaneously.
  * Once the introducer is completely withdrawn, the balloon continues to be inflated until the absence of bleeding is verified.
  * Once hemostasis is achieved, the patient must be able to move his fingers and wrist without bleeding. If bleeding is observed, the balloon is inflated to achieve adequate hemostasis.
  Interventions: Device: Hemostatic device for distal radial approach.
- PreludeSYNC distal (Active Comparator): A specific hemostatic device, designed for distal radial approach.
  * Clean and dry the puncture site.
  * Selection and preparation of the PreludeSYNC distal device according to the approach side.
  * The introducer is withdrawn 2cm.
  * The hemostasis device is placed on the patient's hand.
  * Bands position: 1) little finger side; 2) thumb side; 3) between the thumb and the index finger.
  * The circular mark of the balloon is positioned 1cm proximal to the puncture site.
  * Bands are adjusted and fixed.
  * The syringe is filled with 10 ml of air.
  * The balloon of the device is slowly inflated while the introducer is slowly withdrawn simultaneously.
  * Once the introducer is completely withdrawn, the balloon continues to be inflated until the absence of bleeding is verified.
  * Once hemostasis is achieved, the patient must be able to move his fingers and wrist without bleeding. If bleeding is observed, the balloon should be inflated to achieve adequate hemostasis.
  Interventions: Device: Hemostatic device for distal radial approach.

INTERVENTIONS:
Device: Hemostatic device for distal radial approach. — Hemostasis after distal radial approach is done with one of two devices, one of them is designed specifically for the distal radial approach; the other is not but a modified technique with the last one could be helpful.
  Other Names: PreludeSYNC distal; Terumo Radial Band

SUMMARY:
Comparison of PreludeSYNC distal and Modified Terumo Radial Band in patients with distal radial approach.

DETAILED DESCRIPTION:
INTRODUCTION AND BACKGROUND

Distal radial access at the level of the anatomical snuffbox and dorsal region of the hand has currently positioned itself as a viable and safe approach for procedures in interventional cardiology, whether diagnostic, simple, or complex angioplasties. We know that this approach method mainly reduces the occlusion rate of the proximal radial artery, among other advantages; however, we still do not have scientific evidence on the various hemostasis methods for this approach. Practice varies between centers and countries and hemostasis methods vary from an elastic compression bandage to the use of devices manufactured specifically for this approach such as the PreludeSYNC DISTAL or modification of devices manufactured for proximal radial hemostasis such as the TR band. In this clinical trial, we intend to analyze the efficacy and safety of two hemostasis methods in patients who require an interventional procedure (PredludeSYNC DISTAL vs modified TR band), to date, there is no clinical trial that compares these methods face to-face in relation to their efficacy and safety. Retrospective studies indicate that both methods are effective in reducing radial artery occlusion and are safe in reducing the bleeding/hematoma rate.

THE PURPOSE OF THE STUDY To compare the efficacy (distal radial artery occlusion) and safety (hematoma/bleeding) of two devices of distal radial hemostasis (PreludeSYNC distal and TR band) in patients undergoing percutaneous coronary intervention.

STUDY DESIGN Experimental, randomized, prospective, longitudinal, prolective, and comparative.

SUBJECTS OF STUDY Patients from the Ignacio Chávez National Institute of Cardiology who will undergo distal radial percutaneous coronary intervention/angiography.

METHODOLOGY After signing the informed consent, patients will be randomized by balanced block methods to: 1) Hemostasis using the PreludeSYNC distal device, or 2) Hemostasis using the Modified Radial Band device.

PRIMARY OUTCOME To compare the efficacy (distal radial artery occlusion) and safety (hematoma/bleeding) of PreludeSYNC distal versus Modified Terumo Radial Band in distal radial approach.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease including chronic coronary syndrome or acute coronary syndrome.
* Cardiovascular disease that requires coronary angiography in its approach.

Exclusion Criteria:

* Cardiogenic shock.
* Lesions in venous or arterial hemoducts.
* Impossibility to provide informed consent.
* Chronic kidney disease on hemodialysis through arteriovenous fistula at the same site where the approach is planned.
* Severe chronic renal failure (GFR less than 30 ml/min/m2)
* Patients diagnosed with cancer.
* Patient with rheumatological and hematological pro-thrombotic disorders.
* Non-hydrophilic radial introducer.
* Failed cannulation of the radial artery with an introducer.
* Successful trans-radial access that is crossed over to the femoral approach.
* Patients with an interventional procedure using a radial approach in the previous 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 482 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
To compare the incidence of proximal radial artery occlusion assessed by ultrasound and the incidence of hematoma/bleeding assessed clinically by EASY scale of PreludeSYNC distal versus Modified Terumo Radial Band in distal radial approach. | 24 hours after the procedure. Patients with radial occlusion at 24 hours will be follow at 30 days.
  At 24 hours after the procedure, patients will be evaluated by interrogation, physical exam and ultrasonography. The absence of Doppler flow in the proximal radial artery at wrist level will define the occlusion of the radial artery. The EASY scale will be used to classify the severity of the hematoma in degrees from I to V according to the extension.

SECONDARY OUTCOMES:
Incidence of distal and proximal radial artery occlusion at 24 hours after the procedure. | 24 hours after the procedure.
  Evaluated by clinical signs and doppler.
Radial arterial patency at 30 days in patients with obstruction at 24 hours. | 30 days after the procedure
  Evaluated by clinical signs and ultrasound doppler.
Incidence of hematoma at the approach site. | 24 hours after the procedure.
  Evaluated by clinical signs. Classified according to EASY scale.
Bleeding at the access site. | 24 hours after the procedure.
  Evaluated by clinical signs.
Neurological sequelae. | 24 hours after the procedure.
  Evaluated by clinical signs.
Incidence of radial artery pseudoaneurysms. | 24 hours after the procedure.
  Evaluated by clinical signs and ultrasound doppler.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cardiologia Ignacio Chávez, Mexico City, Mexico